CLINICAL TRIAL: NCT01801254
Title: Using EEG Operant Conditioning to Improve Trait Self-Control and Promote Healthy Behavior
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jordan Silberman, Medical Student, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSRB00043988
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Type II Diabetes; Cardiovascular Disease; Health Behavior
Keywords: Obesity; Type II diabetes; Cardiovascular disease; Health behavior promotion; Neuroeconomics; EEG biofeedback; Low-resolution electromagnetic tomography (LORETA); EEG
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- STRIDES (Experimental): Brain-computer interface training protocol designed to up-regulate specific types of neural activity in regions including the left dorsolateral prefrontal cortex, the anterior cingulate cortex, and Brodmann area 6 bilaterally. Targeted neural activity types are positively associated with self-controlled behavior.
  Interventions: Other: STRIDES
- Sham Control (Sham Comparator): Brain-computer interface training protocol that is designed to have no effect on self-controlled behavior. Stimuli used and durations of training sessions for this protocol are identical to those used in the treatment condition.
  Interventions: Other: Sham Control

INTERVENTIONS:
Other: STRIDES — Self-Control TRaining for Increasing Delay of gratification through EEG operant conditioning with Source localization (STRIDES). Brain-computer interface training protocol designed to up-regulate specific types of neural activity, in regions including the left dorsolateral prefrontal cortex, the anterior cingulate cortex, and Brodmann area 6 bilaterally. Targeted neural activity types are positively associated with self-controlled behavior.
  Arms: STRIDES
Other: Sham Control — Brain-computer interface training protocol that is designed to have no effect on self-controlled behavior.
  Arms: Sham Control

SUMMARY:
The field of neuroeconomics has begun to elucidate neural mechanisms underlying self-control; however, researchers have not yet harnessed neuroeconomics findings to develop interventions for improving self-control ability. The investigators are currently developing such an intervention. The investigators' approach involves using a brain-computer interface with audiovisual feedback to show people what is happening in their own brains, in real time. Through this interface, individuals are trained to increase levels of neural activity that may facilitate self-control, which, in turn, may improve the ability to exhibit self-controlled behaviors. This may increase the ability to engage in heath behaviors for which self-control is required (eg, dieting and exercising). The investigators' long-term goal is to create a tool that will help people develop the self-control needed to achieve lasting improvements in health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Can read and write fluently in English
* At least 18 years of age
* Right-handed
* Overweight or obese (BMI > 24.9)
* Currently has a University of Rochester meal plan
* Currently in contemplation or action stages of change with respect to weight loss (measured with the Weight Stages of Change Algorithm; Rossi, Rossi, Velicer, & Prochaska, 1995).

Exclusion Criteria:

* History of diabetes, epilepsy, celiac disease, lactose intolerance, food allergies, veganism, mental illness, or eating disorders
* Currently taking a medication that may have a strong effect on EEG recordings (eg, an antidepressant, stimulant medication, etc.)
* Currently drinks more than 3 cups of coffee per day or roughly equivalent caffeine intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
postprandial blood glucose and triglycerides | 4 times per week for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Silberman, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States